CLINICAL TRIAL: NCT06838507
Title: Incidence, Characterisation and Outcome-relevance of Perioperative SGLT2 Inhibitor Associated Ketoacidosis - A Multicentre Prospective Cohort Study
Brief Title: Incidence, Characterisation and Outcome-relevance of Perioperative SGLT2 Inhibitor Associated Ketoacidosis
Status: Not yet recruiting | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-2935
Record Dates: First submitted 2025-01-17; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-01

CONDITIONS: SGLT2 Inhibitor; Ketoacidosis, Eugylcemic
MeSH Terms: conditions — Ketosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
The goal of this observational study is to generate data on the incidence and outcome-relevance of sodium-glucose cotransporter 2 (SGLT2) inhibitor associated ketoacidosis in adult patients with regular intake of any SGLT2 inhibitor within the last three months that are undergoing in-patient surgery. Further, it will describe strategies in current clinical practice to prevent and manage SGLT2 inhibitor associated ketoacidosis. The specific aims of this study are:

1. To assess the incidence of SGLT2 inhibitor associated ketoacidosis in surgical patients
2. To characterise fasting times in patients with SGLT2 inhibitor associated ketoacidosis
3. To describe the management of SGLT2 inhibitor associated ketoacidosis in current clinical practice
4. To assess the outcome impact of SGLT2 inhibitor associated ketoacidosis

ELIGIBILITY:
Inclusion Criteria:

* Prescription and regular intakte of any SGLT2 inhibitor within the last three months (regardless if SGLT2 inhibitor was discontinued preoperatively or not)
* Surgical procedure
* At least one overnight stay in the hospital following surgery
* Age >= 18 years

Exclusion Criteria:

* Unwilling and/or unable to consent
* Outpatient surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We aim to recruit patients at 20 German tertiary care centres. Coordinating centre will be the University Hospital Duesseldorf in Duesseldorf.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with postoperative ketoacidosis | From the immediate postoperative period to the first postoperative morning
  Ketoacidosis will be defined as by the American Diabetes Association:
  * pH <= 7,30
  * Serum bicarbonate <= 18 mmol/l
  * Serum and/or urine ketones positive

SECONDARY OUTCOMES:
Composite of postoperative complications | From enrollment to the end of follow up at 30 days after discharge
  Composite of all-cause death, hospital readmission, major adverse cardiovascular events (defined as myocardial infarction, myocardial injury, cardiovascular death, non-fatal cardiac arrest, decompensated heart failure with the need for transfer to a higher unit of care, atrial fibrillation, pulmonary embolism, coronary revascularization), acute kidney injury according to KDIGO criteria or other major postoperative complications (defined as Clavien-Dindo class ≥ 3)
Single postoperative complication | From enrollment to the end of follow up at 30 days after discharge
  Individual components of the composite (all-cause death, hospital readmission, major adverse cardiovascular events (defined as myocardial infarction, myocardial injury, cardiovascular death, non-fatal cardiac arrest, decompensated heart failure with the need for transfer to a higher unit of care, atrial fibrillation, pulmonary embolism, coronary revascularization), acute kidney injury according to KDIGO criteria or other major postoperative complications (defined as Clavien-Dindo class ≥ 3))
Acute kidney injury | From enrollment to the end of follow up at 30 days after discharge
  According to KDIGO definition and based on routinely measured creatinine
Length of stay in-hospital | From enrollment to discharge (in-hospital) at approximately four days after surgery
Length of stay on intensive care unit | From entering the intensive care unit to discharge to the normal ward at approximately 2 days after surgery
Length of stay in the recovery room | From entering the recovery room to discharge to the normal ward at approximately one hour after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesiology, University Hospital Duesseldorf, Düsseldorf, Germany

REFERENCES:
- [Background] Lurati Buse GA, Mauermann E, Ionescu D, Szczeklik W, De Hert S, Filipovic M, Beck-Schimmer B, Spadaro S, Matute P, Bolliger D, Turhan SC, van Waes J, Lagarto F, Theodoraki K, Gupta A, Gillmann HJ, Guzzetti L, Kotfis K, Wulf H, Larmann J, Corneci D, Chammartin-Basnet F, Howell SJ; MET: Reevaluation for Perioperative Cardiac Risk investigators; European Society of Anaesthesiology and Intensive Care. Risk assessment for major adverse cardiovascular events after noncardiac surgery using self-reported functional capacity: international prospective cohort study. Br J Anaesth. 2023 Jun;130(6):655-665. doi: 10.1016/j.bja.2023.02.030. Epub 2023 Apr 1. PMID 37012173
- [Background] Steinhorn B, Wiener-Kronish J. Dose-dependent relationship between SGLT2 inhibitor hold time and risk for postoperative anion gap acidosis: a single-centre retrospective analysis. Br J Anaesth. 2023 Oct;131(4):682-686. doi: 10.1016/j.bja.2023.06.063. Epub 2023 Aug 2. PMID 37541949
- [Background] Ruste M, Schweizer R, Groisne L, Fellahi JL, Jacquet-Lagreze M. Sodium-glucose cotransporter-2 inhibitors in non-diabetic patients: is there a perioperative risk of euglycaemic ketoacidosis. Br J Anaesth. 2024 Feb;132(2):435-436. doi: 10.1016/j.bja.2023.11.015. Epub 2023 Dec 4. No abstract available. PMID 38052677
- [Background] Oosterom-Eijmael MJP, Hermanides J, van Raalte DH, Hulst AH. Risk of perioperative discontinuation of SGLT2 inhibitors. Br J Anaesth. 2024 Aug;133(2):239-240. doi: 10.1016/j.bja.2024.05.004. Epub 2024 Jun 4. PMID 38834489
- [Background] Thiruvenkatarajan V, Meyer EJ, Nanjappa N, Van Wijk RM, Jesudason D. Perioperative diabetic ketoacidosis associated with sodium-glucose co-transporter-2 inhibitors: a systematic review. Br J Anaesth. 2019 Jul;123(1):27-36. doi: 10.1016/j.bja.2019.03.028. Epub 2019 May 3. PMID 31060732
- [Background] Colacci M, Fralick J, Odutayo A, Fralick M. Sodium-Glucose Cotransporter-2 Inhibitors and Risk of Diabetic Ketoacidosis Among Adults With Type 2 Diabetes: A Systematic Review and Meta-Analysis. Can J Diabetes. 2022 Feb;46(1):10-15.e2. doi: 10.1016/j.jcjd.2021.04.006. Epub 2021 Apr 28. PMID 34116926
- [Background] Long B, Lentz S, Koyfman A, Gottlieb M. Euglycemic diabetic ketoacidosis: Etiologies, evaluation, and management. Am J Emerg Med. 2021 Jun;44:157-160. doi: 10.1016/j.ajem.2021.02.015. Epub 2021 Feb 16. PMID 33626481
- [Background] Musso G, Saba F, Cassader M, Gambino R. Diabetic ketoacidosis with SGLT2 inhibitors. BMJ. 2020 Nov 12;371:m4147. doi: 10.1136/bmj.m4147. No abstract available. PMID 33184044
- [Background] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Skibelund AK; ESC Scientific Document Group. 2023 Focused Update of the 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2023 Oct 1;44(37):3627-3639. doi: 10.1093/eurheartj/ehad195. No abstract available. PMID 37622666
- [Background] Nuffield Department of Population Health Renal Studies Group; SGLT2 inhibitor Meta-Analysis Cardio-Renal Trialists' Consortium. Impact of diabetes on the effects of sodium glucose co-transporter-2 inhibitors on kidney outcomes: collaborative meta-analysis of large placebo-controlled trials. Lancet. 2022 Nov 19;400(10365):1788-1801. doi: 10.1016/S0140-6736(22)02074-8. Epub 2022 Nov 6. PMID 36351458
- [Background] Solomon SD, McMurray JJV, Claggett B, de Boer RA, DeMets D, Hernandez AF, Inzucchi SE, Kosiborod MN, Lam CSP, Martinez F, Shah SJ, Desai AS, Jhund PS, Belohlavek J, Chiang CE, Borleffs CJW, Comin-Colet J, Dobreanu D, Drozdz J, Fang JC, Alcocer-Gamba MA, Al Habeeb W, Han Y, Cabrera Honorio JW, Janssens SP, Katova T, Kitakaze M, Merkely B, O'Meara E, Saraiva JFK, Tereshchenko SN, Thierer J, Vaduganathan M, Vardeny O, Verma S, Pham VN, Wilderang U, Zaozerska N, Bachus E, Lindholm D, Petersson M, Langkilde AM; DELIVER Trial Committees and Investigators. Dapagliflozin in Heart Failure with Mildly Reduced or Preserved Ejection Fraction. N Engl J Med. 2022 Sep 22;387(12):1089-1098. doi: 10.1056/NEJMoa2206286. Epub 2022 Aug 27. PMID 36027570
- [Background] McMurray JJV, Solomon SD, Inzucchi SE, Kober L, Kosiborod MN, Martinez FA, Ponikowski P, Sabatine MS, Anand IS, Belohlavek J, Bohm M, Chiang CE, Chopra VK, de Boer RA, Desai AS, Diez M, Drozdz J, Dukat A, Ge J, Howlett JG, Katova T, Kitakaze M, Ljungman CEA, Merkely B, Nicolau JC, O'Meara E, Petrie MC, Vinh PN, Schou M, Tereshchenko S, Verma S, Held C, DeMets DL, Docherty KF, Jhund PS, Bengtsson O, Sjostrand M, Langkilde AM; DAPA-HF Trial Committees and Investigators. Dapagliflozin in Patients with Heart Failure and Reduced Ejection Fraction. N Engl J Med. 2019 Nov 21;381(21):1995-2008. doi: 10.1056/NEJMoa1911303. Epub 2019 Sep 19. PMID 31535829
- [Background] Zinman B, Wanner C, Lachin JM, Fitchett D, Bluhmki E, Hantel S, Mattheus M, Devins T, Johansen OE, Woerle HJ, Broedl UC, Inzucchi SE; EMPA-REG OUTCOME Investigators. Empagliflozin, Cardiovascular Outcomes, and Mortality in Type 2 Diabetes. N Engl J Med. 2015 Nov 26;373(22):2117-28. doi: 10.1056/NEJMoa1504720. Epub 2015 Sep 17. PMID 26378978